CLINICAL TRIAL: NCT00568100
Title: Effect of Pressure Support Ventilation and Neurally Adjusted Ventilatory Assist (NAVA) in COPD Patients
Brief Title: Effect of Pressure Support Ventilation and Neurally Adjusted Ventilatory Assist (NAVA) in Chronic Obstructive Pulmonary Disease (COPD) Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Policlinico Hospital (Other)
Responsible Party: Principal Investigator, Davide Chiumello, MD, Policlinico Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2222
Record Dates: First submitted 2007-12-04; First posted 2007-12-05 (Estimated); Last update posted 2015-04-28 (Estimated); Status verified 2015-04

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: gas exchange; pressure support ventilation; respiratory mechanics; COPD; NAVA
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): COPD patients
  Interventions: Procedure: PSV and NAVA

INTERVENTIONS:
Procedure: PSV and NAVA — evaluated the effect of PSV and NAVA on breathing pattern, respiratory effort, gas exchange and level of breathing comfort in COPD patients

SUMMARY:
The investigators' aim is to study the effect of pressure support ventilation at two levels of PEEP and Pressure Support versus neurally adjusted ventilatory assist (NAVA) in COPD patients.

DETAILED DESCRIPTION:
In this study, two levels of pressure support and PEEP during pressure support ventilation are compared with neurally adjusted ventilatory assist (NAVA) in COPD patients by measuring respiratory mechanics, intrinsic PEEP, work of breathing and patient's level of comfort.

ELIGIBILITY:
Inclusion Criteria:

* Stable COPD patients during non invasive mechanical ventilation

Exclusion Criteria:

* Haemodynamic instability
* Coma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2010-04; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Respiratory mechanics, gas exchange, work of breathing | 5 minutes

SECONDARY OUTCOMES:
Comfort of breathing | 5 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Davide Chiumello, MD, Principal Investigator — Policlinico Hospital
Locations (1):
- Policlinico Hospital, Milan, Italy